




# Statistical Analysis Plan

A Randomized Multicenter Study of Ibrutinib in Combination with Pomalidomide and Dexamethasone in Subjects with Relapsed/Refractory Multiple Myeloma

**PCYC-1138-CA** 

June 26, 2018

Version 2.0

The information in this document is considered privileged and confidential by Pharmacyclics LLC, and may not be disclosed to others except to the extent necessary to obtain Institutional Review Board approval and informed consent, or as required by Federal and State Laws. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed.

opharmacyclics An Abbitic Company

# PCYC-1138-CA

Statistical Analysis Plan


## Statistical Analysis Plan Approval

| TIOUSCOLINGIIISCI. | Protocol | Number: |
|--------------------|----------|---------|
|--------------------|----------|---------|

PCYC-1138-CA

Protocol Title:

A Randomized Multicenter Study of Ibrutinib in Combination

with Pomalidomide and Dexamethasone in Subjects with

Relapsed/Refractory Multiple Myeloma

SAP Version:

2.0

Date:

26JUN2018

By signing below, all parties accept that the analysis methods and data presentations are acceptable and that this document is final.

| acceptable and that this document is final. | |
|---|---|
| Yihua Lee, PhD Associate Director, Biostatistics | D9- JUL-2018 Date (ddMMMyyyy) |
| Edyta Dobkowska, MD<br>Medical Director, Clinical Science | Date (ddMMMyyyy) |
| Thorsten Graef, MD, PhD Head of Clinical Development | Date (ddMMMyyyy) |
| Claire Tsao, PhD<br>Senior Director, Biostatistics | Date (ddMMMyyyy) |
| Andreas Terjung Senior Director, Regulatory Affairs | Date (ddMMMyyyy) |
| Harnisha Dalwadi, PhD<br>Senior Director, Medical Writing | Date (ddMMMyyyy) |




## Statistical Analysis Plan Approva

| 38-C# |
|-------|

Protocol Title: A Randomized Multicenter Study of Ibrutinib in Combination

with Pomalidomide and Dexamethasone in Subjects with

Relapsed/Refractory Multiple Myeloma

SAP Version: 2.0

Date: 26JUN2018

By signing below, all parties accept that the analysis methods and data presentations are acceptable and that this document is final.

| Vihua Lee, PhD | Date (ddMMMyyyy) |
|-------------------------------------|-------------------------|
| Associate Director, Biostatistics | |
| 0. | |
| Totale Dellowska | S3 JANE 5018 |
| Edyta Dobkowska, MD | Date (ddMMMyyyy) |
| Medical Director, Clinical Science | |
| Thorsten Graef, MD | Date (ddMMMyyyy) |
| Head of Oncology | Date (delivityliggy) |
| Claire Tsao, PhD | Date (ddMMMyyyy) |
| Senior Director, Biostatistics | Date (delivitylitylyyy) |
| Andreas Terjung | Date (ddMMMyyyy) |
| Senior Director, Regulatory Affairs | |
| Harnisha Dalwadi, PhD | Date (ddMMMyyyy) |
| Senior Director, Medical Writing | ( |




## Statistical Analysis Plan Approval

| Protocol Number: | PCYC-1138-CA | Λ | |
|---|---|---|---|
| Protocol Title: | with Pomalidon | A Randomized Multicenter Study of Ibrutinib in Combination with Pomalidomide and Dexamethasone in Subjects with Relapsed/Refractory Multiple Myeloma | |
| SAP Version: | 2.0 | | |
| Date: | 26JUN2018 | | |
| By signing below, all parties acceptable and that this docu | _ | lysis methods and data presentations | are |
| Yihua Lee, PhD<br>Associate Director, Biostatis | stics | Date (ddMMMyyyy) | |
| Edyta Dobkowska, MD<br>Medical Director, Chinical S | cience | Date (ddMMMyyyy) | |
| 1 | | Date (ddMMMyyyy) | |
| Thorsten Graef, MD, PhD<br>Head of Clinical Developme | ent | Date (ddMMMyyyy) | |
| Claire Tsao, PhD<br>Senior Director, Biostatistics | S | Date (ddMMMyyyy) | |
| Andreas Terjung Senior Director, Regulatory | Affairs | Date (ddMMMyyyy) | |
| Harnisha Dalwadi, PhD | | Date (ddMMMyyyy) | - |

Senior Director, Medical Writing




# **Statistical Analysis Plan Approval**

| Protocol Number: | PCYC-1138- | CA |
|---|---|---|
| with Pomalido | | ed Multicenter Study of Ibrutinib in Combination lomide and Dexamethasone in Subjects with fractory Multiple Myeloma |
| SAP Version: | 2.0 | |
| Date: | 26JUN2018 | |
| By signing below, all partinceptable and that this do | • | analysis methods and data presentations are |
| Yihua Lee, PhD<br>Associate Director, Biosta | tistics | Date (ddMMMyyyy) |
| Edyta Dobkowska, MD<br>Medical Director, Clinical | Science | Date (ddMMMyyyy) |
| Thorsten Graef, MD<br>Head of Oncology | | Date (ddMMMyyyy) |
| Claire Tsao, PhD<br>Senior Director, Biostatist | ics | 26Jun2018 Date (ddMMMyyyy) |
| Andreas Terjung<br>Senior Director, Regulator | ry Affairs | Date (ddMMMyyyy) |
| Harnisha Dalwadi, PhD<br>Senior Director, Medical V | Writing | Date (ddMMMyyyy) |




# Statistical Analysis Plan Approval

| Protocol Number: PCYC-1138-CA | |
|---|---|
| Protocol Title: | A Randomized Multicenter Study of Ibrutinib in Combination with Pomalidomide and Dexamethasone in Subjects with Relapsed/Refractory Multiple Myeloma |
| SAP Version: | 2.0 |
| Date: | 26JUN2018 |
| By signing below, all parties a acceptable and that this documents | eccept that the analysis methods and data presentations are ent is final. |
| Yihua Lee, PhD<br>Associate Director, Biostatisti | Date (ddMMMyyyy) |
| Edyta Dobkowska, MD<br>Medical Director, Clinical Sci | Date (ddMMMyyyy) |
| Thorsten Graef, MD<br>Head of Oncology | Date (ddMMMyyyy) |
| Claire Tsao, PhD<br>Senior Director, Biostatistics | Date (ddMMMyyyy) |
| Andreas Terjung Senior Director, Regulatory A | Date (ddMMMyyyy) Ffairs |
| Harnisha Dalwadi, PhD<br>Senior Director, Medical Writ | Date (ddMMMyyyy) |




# **Statistical Analysis Plan Approval**

| Protocol Number: | PCYC-1138-CA |
|---|---|
| Protocol Title: | A Randomized Multicenter Study of Ibrutinib in Combination with Pomalidomide and Dexamethasone in Subjects with Relapsed/Refractory Multiple Myeloma |
| SAP Version: | 2.0 |
| Date: | 26JUN2018 |
| By signing below, all parties a acceptable and that this document | accept that the analysis methods and data presentations are nent is final. |
| Yihua Lee, PhD<br>Associate Director, Biostatisti | Date (ddMMMyyyy) |
| Edyta Dobkowska, MD<br>Medical Director, Clinical Sci | Date (ddMMMyyyy) |
| Thorsten Graef, MD<br>Head of Oncology | Date (ddMMMyyyy) |
| Claire Tsao, PhD<br>Senior Director, Biostatistics | Date (ddMMMyyyy) |
| Andreas Terjung<br>Senior Director, Regulatory A | Date (ddMMMyyyy) |
| HANLMAN | 29 June 2018 |
| Harnisha Dalwadi, PhD | Date (ddMMMyyyy) |




## **TABLE OF CONTENTS**

| LI | ST O | OF ABBREVIATIONS | 4 |
|----|------|-------------------------------------------|----|
| 1 | INT | TRODUCTION | 5 |
| | 1.1 | Study Design – Phase 1 | |
| | 1.2 | Objective/Endpoints of Study – Phase 1 | 6 |
| | | Primary Objective | 6 |
| | | Secondary Endpoints | 6 |
| | 1.3 | Sample Size Determination | 6 |
| | 1.4 | Planned Analysis | 6 |
| | | Final Analysis | 6 |
| 2 | GE | NERAL ANALYSIS CONSIDERATION | 6 |
| | 2.1 | Analysis Sets | |
| 3 | SUE | BJECT INFORMATION | 8 |
| | 3.1 | Subject Disposition | |
| | 3.2 | Demographics and Baseline Characteristics | |
| | 3.3 | Concomitant Medications | 8 |
| | 3.4 | Extent of Exposure to Study Treatment | 8 |
| 4 | AN | ALYSIS FOR ENDPOINTS | 9 |
| 5 | SAI | FETY ASSESSMENTS | 10 |
| 6 | CH | ANGES IN PROTOCOL PLANNED ANALYSIS | |
| 7 | REI | FERENCES | 12 |




#### LIST OF ABBREVIATIONS

AE adverse event

ATC Anatomical Therapeutic Chemical

CBR clinical benefit rate
CI confidence interval
CR complete response
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DCB Duration of Clinical Benefit
DOR duration of overall response

Hgb hemoglobin

MedDRA Medical Dictionary for Regulatory Activities

MR minimal response

NCI National Cancer Institute
ORR overall response rate

PCYC Pharmacyclics
PD progressive disease
PR partial response
PT preferred term

SAP statistical analysis plan

TEAE treatment-emergent adverse events

#### 1 INTRODUCTION

The Study PCYC-1138-CA consisted of a Phase 1 and a Phase 2 part. After completion of the Phase 1 part, in which 11 subjects received study treatment, the sponsor decided to not pursue an indication for treatment of patients with multiple myeloma with ibrutinib and therefore terminate the study early. Thus, this statistical analysis plan (SAP) is to define only the key study elements for the Phase 1 part of the study including variable definitions, and statistical methods for analysis of data in evaluation of efficacy and safety. Analyses of pharmacokinetics data will be addressed in a separate document. Biomarker analysis will not be performed due to early termination of the study. Throughout this SAP, "study treatment" and "study drug" are used interchangeably.

Analysis methods specified in this document take precedence over those described in the study protocol should there be any difference.

#### 1.1 Study Design – Phase 1

The Phase 1 part of the study was an open-label, international, multicenter dose-finding study of the ibrutinib, pomalidomide and dexamethasone combination in subjects with relapsed/refractory multiple myeloma (MM). Up to 18 patients were to be enrolled in order to determine the maximum therapeutic dose/maximum administered dose (MTD/MAD). In the dose finding portion of the study, up to 2 cohorts were to be explored (Table 1). The study followed a 3+3+3 dose escalation design. The MTD/MAD was defined as the highest dose level at which <33% (ie,  $\le 1$  of 6 or  $\le 2$  of 9) of subjects in a cohort experience a study treatment related dose limiting toxicity (DLT).

**Table 1: Dosing Levels and Cohorts** 

| Dose Level | Cohort | Ibrutinib <sup>a</sup> | Pomalidomide <sup>b</sup> | <b>Dexamethasone</b> <sup>c</sup> |
|---|---|---|---|---|
| -1 | -1 | 420 mg once daily | 4 mg | 40 mg |
| 1 (Starting Dose) | 1 | 560 mg once daily | 4 mg | 40 mg |
| 2 | 2 | 840 mg once daily | 4 mg | 40 mg |

<sup>&</sup>lt;sup>a.</sup> Ibrutinib was administered PO starting on Day 1 of Cycle 1, dosing was continuous thereafter (without interruption).

b. Pomalidomide was administered PO on Days 1 – 21 of a 28-day cycle.

<sup>&</sup>lt;sup>c.</sup> Dexamethasone was administered PO once weekly. The dose was reduced to 20 mg weekly in those >75 years of age


### 1.2 Objective/Endpoints of Study – Phase 1

### • Primary Objective

- o To determine the MTD)/ MAD of the ibrutinib, pomalidomide and dexamethasone combination.
- To determine the safety and tolerability of ibrutinib in combination with pomalidomide and dexamethasone in subjects with relapsed/refractory MM.

### • Secondary Endpoints

- Overall response rate (ORR): partial response (PR) or better, per the International Myeloma Working Group (IMWG) response criteria (Rajkumar 2011)<sup>1,2,3</sup>
- o Duration of Response (DOR)
- o The clinical benefit rate (CBR) and its duration, defined as ≥ minimal response (MR) according to the IMWG response criteria
- o To evaluate the pharmacokinetics (PK) of ibrutinib and pomalidomide when given in combination with dexamethasone

#### 1.3 Sample Size Determination

Phase 1: This was a standard 3+3+3 design to determine the MTD/MAD and toxicity profile of ibrutinib in combination with pomalidomide and dexamethasone. Dose escalation were to follow the 3+3+3 principle and up to 2 cohorts were to be explored. This study was not powered for comparison of treatment cohorts. Up to 18 subjects were to be enrolled into the Phase 1 part of the study.

#### 1.4 Planned Analysis

#### • Final Analysis

The final analysis for the clinical study report will be conducted when all Phase 1 subjects have exited PCYC-1138-CA study. The sponsor decided not to perform the Phase 2 part of the study following a decision not to pursue an indication for multiple myeloma for ibrutinib.

#### 2 GENERAL ANALYSIS CONSIDERATION

Subjects will be analyzed and summarized for safety and other selected endpoints.

#### 2.1 Analysis Sets

#### Safety Population

The safety population include subjects who have received any dose of study treatment.




### o Response-Evaluable Population

The response-evaluable population is defined as subjects who are in safety population and provided at least one post-baseline response (or disease) assessment. All subjects in safety population received at least 1 post-baseline response assessment.


#### 3 SUBJECT INFORMATION

### 3.1 Subject Disposition

The disposition tables will include the following summaries.

- Analysis population
- Study Treatment Disposition and Discontinuation
- Study Status, Duration of Treatment and Study Exit

Time on study is defined as the interval between the date of first dose and the date of last known to have been alive. The Kaplan-Meier method will be used to estimate the median time on study with subjects who died being censored at death date.

### 3.2 Demographics and Baseline Characteristics

Subject demographics, baseline characteristics and baseline disease characteristics will be summarized with descriptive statistics for the safety population.

#### 3.3 Concomitant Medications

Medications will be coded to Anatomical Therapeutic Chemical (ATC) class and the preferred drug name (hereafter referred as "preferred name") per World Health Organization drug dictionary. Listings will be provided to present the data.

Concomitant CYP3A inhibitors and inducers taken any time while on study treatment (i.e., from the date of first dose through the date of last dose of the study treatment) will be summarized by ATC class and preferred term (PT). Each subject will be counted once for each PT, and each ATC class.

### 3.4 Extent of Exposure to Study Treatment

Exposure to the 3 study drugs will be summarized for the safety population. Descriptive statistics will be provided for the following data for each of the 3 drugs unless otherwise specified: treatment duration (month) and number (%) of subjects with dose reduction due to adverse events (AEs).


### **ANALYSIS FOR ENDPOINTS**

Analysis of secondary endpoints (Table 2) will be conducted on the safety population.

**Table 2: Definitions and Analyses for Secondary Endpoints** 

| Endpoint | Definition | Analysis Method |
|---|---|---|
| Secondary endpoints: | | |
| Overall Response<br>Rate (ORR) | The proportion of subjects achieving a best overall response of PR or better per investigator assessment per IMWG at or prior to initiation of subsequent anticancer therapy | ORR will be estimated and the corresponding 2-sided 95% exact binomial confidence interval will be calculated. |
| Duration of<br>Response (DOR) | The time interval between the date of initial documentation of a response and the date of first documented evidence of PD, death, or date of censoring for the subjects not progressed/died. The censoring date is the last adequate tumor assessment date. | A listing will be provided. |
| Clinical Benefit<br>Rate (CBR) | The proportion of subjects achieving a best overall response of MR or better per investigator assessment per IMWG at or prior to initiation of subsequent anticancer therapy | CBR will be estimated and the corresponding 2-sided 95% exact binomial confidence interval will be calculated. |

Note: DOR; duration of response; PD: disease progression; PR: partial response; MR: minimal response;

IMWG: International Myeloma Working Group.


### 5 <u>SAFETY ASSESSMENTS</u>

Safety data will be summarized for safety population unless otherwise indicated. Table 3 summarizes the safety analyses to be carried out. AEs will be coded in accordance with the Medical Dictionary for Regulatory Activities (MedDRA). Severity of AEs were graded by the investigator according the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03. A listing will be provided to indicate dose-limiting toxicity (DLT).

In general, the treatment-emergent period is defined as the period from the date of the first dose of study treatment up to 30 days after the date of the last dose of study treatment or the day before initiation of subsequent anticancer therapy, whichever comes first. Treatment emergent AEs are those events that occur or worsen during the treatment-emergent period or that are related to the study treatment or events with a complete missing onset date but with a resolution date during the treatment phase.

All laboratory values will be converted to and reported as international standard (SI) units. In general, only data from the central laboratory will be summarized and analyzed. Laboratory parameters will be graded using the NCI CTCAE v4.03.

**Table 3: Summary of Safety Assessments** 

| Assessment Type | Definition | Analysis Methods |
|---|---|---|
| AE | TEAEs, SAEs, non-serious TEAE, grade 3 or worse TEAEs, related TEAEs, TEAEs leading to treatment discontinuation, TEAEs leading to dose reduction, TEAEs leading to death, protocol- defined events of special interest and other safety observations | Descriptive summary statistics and/or listings |
| Lab | Worst post-baseline toxicity grade for selected CTCAE gradable hematology and chemistry. Abnormalities in creatinine clearance, uric acid, and liver function | Descriptive summary statistics and/or listings |
| Vital Signs and other<br>Observations Related to<br>Safety | SBP, DBP, weight, heart rate, new or worsened eye-related symptoms | Descriptive summary statistics and/or listings |
| Dose Limiting Toxicity (DLT) | DLT | Listing |

TEAE: treatment-emergent adverse event; SAE= serious adverse event; SBP: systolic blood pressure; DBP: diastolic blood pressure; CTCAE= Common Terminology Criteria for Adverse Events.




#### 6 CHANGES IN PROTOCOL PLANNED ANALYSIS

The following modifications to the protocol "Statistical Methods and Analysis" section is made due to the decision by sponsor to terminate the study early.

- 1) Phase 2 part of the study was not initiated, therefore, the analysis for Phase 2 will not be performed.
- 2) Biomarker analysis will not be performed due to early termination of the study.
- 3) The secondary endpoint of the duration of clinical benefit response will not be performed due to the early termination of the study.




#### 7 REFERENCES

- 1. Anderson KC, Kyle RA, Rajkumar SV, et al. Clinically relevant end points and new drug approvals for myeloma. Leukemia 2008; 22(2):231-239.
- 2. Durie BG, Harousseau JL, Miguel JS, et al. International uniform response criteria for multiple myeloma. Leukemia 2006; 20(9):1467-1473.
- 3. Rajkumar SV, Harousseau JL, Durie B, et al. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood 2011; 117(18): 4691-4695.